CLINICAL TRIAL: NCT04003324
Title: Users' Experiences and Preliminary Efficacy of a Self-monitoring Tool to Reduce Sedentary Behavior in Older Adults: a Mixed-methods Study
Brief Title: Reducing Older Adults' Sedentary Behavior by Self-monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VakgroepBewegingsEnSportwetenschappen (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor-Investigator, VakgroepBewegingsEnSportwetenschappen, Head of the Department - Prof. Greet Cardon, University Ghent
Organization: University Ghent (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Op is Top - Pilot
Record Dates: First submitted 2019-03-13; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior | interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Self-monitoring tool (Activator) and general information
  Interventions: Behavioral: Op is Top - using feedback from the Activator to reduce sedentary behavior in older adults

INTERVENTIONS:
Behavioral: Op is Top - using feedback from the Activator to reduce sedentary behavior in older adults — Participants will receive a self-monitoring tool (i.e. the Activator) aimed at the reduction of sedentary behavior. Participants will be able to use the self-monitoring tool for four weeks. Apart from that, participants will receive general sedentary behavior information and an explanation on how to use the self-monitoring tool.

SUMMARY:
The first aim of this study is to gain insight into older adults' perceptions towards a self-monitoring tool aimed at the reduction of sedentary behavior. Secondly, this study aimed to investigate the preliminary efficacy of a self-monitoring tool aimed at the reduction of sedentary behavior.

DETAILED DESCRIPTION:
A mixed-method study will be conducted to assess participants' perceptions and preliminary efficacy of a self-monitoring based intervention aimed at the reduction of sedentary behavior in older adults (> 60 years).

A convenience sample of 40 older adults will be recruited using Facebook advertisements, as well as from an existing database of older adults willing to participate in research studies.

Older adults who agree to participate will be contacted by phone to make an appointment for a visit. During this first visit, participants will receive an informed consent. After signing the informed consent, a structured interview will be conducted to assess the participants' socio-demographic characteristics, domain-specific sedentary behavior and health status. A semi-structured interview will be conducted to examine participants' perceptions towards (reducing) sedentary behavior. Moreover, an inclinometer will be attached to the participants' thigh. Participants will be instructed to wear the inclinometer for one week. After one week, a researcher will visit the participants once again to collect the inclinometers. During this second visit, participants will receive a self-monitoring tool (i.e. the Activator) aimed at the reduction of sedentary behavior. Participants will be able to use the self-monitoring tool for four weeks. Apart from that, participants will receive a booklet with general sedentary behavior information and an explanation on how to use the self-monitoring tool. By the end of the intervention, the self-monitoring tools will be collected, and participants will be instructed to answer another structured interview and to wear the inclinometer for another week. At the end of this week, inclinometers will collected, and a semi-structured interview will be conducted with the older adults of the intervention group to gain insight into their experiences with self-monitoring as a behavior change technique to reduce sedentary behavior, as well as with the Activator.

ELIGIBILITY:
Inclusion Criteria:

* be at least 60 years old
* be Dutch-speaking
* be able to walk 100 meters without severe difficulties
* have a smartphone

Exclusion Criteria:

- having functional limitations to stand up

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Total sedentary behavior | Pretest - posttest (4 weeks)
  Total sedentary behavior was objectively estimated by means of the ActivPAL inclinometer (PAL Technologies, Glasgow, UK). The inclinometer was attached on the midline of the right anterior thigh. Participants were instructed to wear the inclinometer for seven consecutive days (24h/day) both at baseline, and at post measurement.
Perceptions of (reducing) sedentary behavior | Posttest (4 weeks)
  Perceptions of older adults' towards reducing sedentary behavior by means of a self-monitoring tool will be assessed using a semi-structured interview. The interview guide has been developed by the principal investigator and includes open questions regarding older adults' perceptions towards 1) sedentary behavior, 2) using self-monitoring to reduce sedentary behavior and 3) the Activator (i.e. the self-monitoring tool used in our study). Examples of questions are: What are your perceptions regarding the Activator? Did you enjoy receiving feedback on your sitting time every day? Etc.
Domain-specific sedentary behavior | Pretest - posttest (4 weeks)
  Domain-specific sedentary behaviors were assessed using a questionnaire developed by Busschaert et al. Concretely, week and weekend day sedentary behaviors were asked using the following question: 'During the last 7 days, how much time did you usually spend sitting while (1) reading, (2) caring, (3) practicing hobbies, (4) socializing, (5) listening to/playing music, (6) consuming meals, (7) watching television, (8) using a computer, (9) moving from one place to another, (10) doing household activities (11) making phone calls.

CONTACTS AND LOCATIONS:
Overall Officials: Greet Cardon, Prof., Study Director — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Compernolle S, Van Dyck D, Cardon G, Brondeel R. Exploring Breaks in Sedentary Behavior of Older Adults Immediately After Receiving Personalized Haptic Feedback: Intervention Study. JMIR Mhealth Uhealth. 2021 May 10;9(5):e26387. doi: 10.2196/26387. PMID 33970109
- [Derived] Compernolle S, Cardon G, van der Ploeg HP, Van Nassau F, De Bourdeaudhuij I, Jelsma JJ, Brondeel R, Van Dyck D. Engagement, Acceptability, Usability, and Preliminary Efficacy of a Self-Monitoring Mobile Health Intervention to Reduce Sedentary Behavior in Belgian Older Adults: Mixed Methods Study. JMIR Mhealth Uhealth. 2020 Oct 29;8(10):e18653. doi: 10.2196/18653. PMID 33118951